CLINICAL TRIAL: NCT06448442
Title: A Pilot Study of Deep Cervical Lymphatic-venous Anastomosis in the Treatment of Alzheimer's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Yuanjian Fang, Dr., Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2024-0429
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Safety Issues; Feasibility; Therapeutic Value

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alzheimer's disease (AD) is the most prevalent form of dementia, affecting 3-4% of the population over a lifetime. It's characterized by abnormal Amyloid-beta (Aβ) and tau protein expression and accumulation in the central nervous system, leading to amyloid plaques and neurofibrillary tangles. While current treatments can slow cognitive decline, there's no cure.

The discovery of the "glymphatic-meningeal lymphatic" system has shed new light on cerebrospinal fluid circulation, showing it has a similar interstitial fluid system to peripheral lymphatic circulation. This system helps clear waste and transport nutrients in the brain, known as the glymphatic phenomenon. The deep cervical lymph nodes, part of this system, are crucial for cerebrospinal fluid drainage and are linked to the clearance of AD-related proteins.

Aging and inflammation can impair deep cervical lymph node function, increasing cerebrospinal fluid drainage pressure and potentially contributing to AD progression. Lymphatic anastomosis, a surgical technique used for lymphedema and other conditions, is being explored as a potential treatment to alleviate neurodegenerative disease by reducing cerebrospinal fluid pressure and clearing metabolic waste.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common form of dementia, with an estimated lifetime prevalence rate of 3-4%. Its characteristics include abnormal expression of Amyloid-beta (Aβ) and tau proteins, as well as their accumulation in the central nervous system. The aggregated toxic proteins further form amyloid plaques and neurofibrillary tangles. One of the biggest scientific and therapeutic challenges of AD is to elucidate this protein pathology and how it leads to accumulation in the central nervous system. Although current drug treatment options can slow down the decline in cognitive abilities, there is no treatment strategy to improve the disease.

Recently, the revelation of the "glymphatic-meningeal lymphatic" system has updated the latest theory of cerebrospinal fluid circulation. There is an interstitial fluid circulation system in the brain tissue that is similar to peripheral lymphatic circulation. Research has found that cerebrospinal fluid in the brain enters the perivascular space around the veins through the perivascular space around the arteries, directed by the astrocyte Aquaporin protein-4, which promotes the clearance of waste and the transport of nutrients in the brain, a phenomenon known as the glymphatic phenomenon. At the same time, research has found that there are a large number of lymphatic vessels on both sides of the dural venous sinuses, which participate in the drainage of cerebrospinal fluid and eventually converge into the deep cervical lymph nodes. In animal models of AD and Parkinson's disease (PD), the "glymphatic-meningeal lymphatic" drainage function is significantly related to the clearance of disease-related proteins such as amyloid beta (Aβ), tau, and alpha-synuclein. Ligation of the deep cervical lymph nodes significantly exacerbates the progression of the disease. At the same time, clinical studies have confirmed the decline of "glymphatic-meningeal lymphatic" function in patients with AD and PD through magnetic resonance imaging technology.

The deep cervical lymph nodes play an important role as the final destination of cerebrospinal fluid drainage in the "glymphatic-cranial lymphatic" system. With aging, infection, and chronic inflammation, the function of the deep cervical lymph nodes gradually declines, which will significantly increase the pressure of cerebrospinal fluid circulation and reflux in the brain. The large amount of neurotoxic substances produced during the progression of AD, will further lead to the dysfunction of the deep cervical lymph nodes, ultimately leading to abnormal accumulation of toxic substances in the brain and the progression of the disease. Lymphatic anastomosis is a surgical technique widely used for limb lymphedema, post-traumatic chylous chest, breast cancer, and other post-tumor resection local edema and other diseases, with high safety, reliability, and ease of operation, and has been proven to have many advantages after half a century of testing. Currently, many hospitals at home and abroad have carried out related operations, all of which have achieved good results. Recently, only in our province, Zhejiang Provincial People's Hospital, Taizhou Hospital, Hangzhou Qiushi Hospital, and others have carried out related operations, and the famous Cleveland Clinic in the United States is also conducting related surgical treatment research.

We speculate that anastomosing the corresponding lymphatic vessels in the neck with the veins (Deep Cervical Lymph-Venous anastomosis) might reduce the cerebrospinal fluid circulation pressure in the brain tissue, accelerate the return of interstitial fluid in the brain tissue, clear the accumulation of metabolic products, and alleviate the progression of neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* a. aged 50-90 years (> or equal to 50 years old, < or equal to 90 years old) were evaluated as Alzheimer's disease group according to the 2018 NIA-AA diagnostic criteria; B. signed by the patient or family informed consent; c. Patients with mild or moderate disease, 11≤MMSE≤26; d. Subjects with primary school education or above can complete the prescribed scale evaluation; The diagnosis of AD was confirmed by e.PET or cerebrospinal fluid examination

Exclusion Criteria:

* a. any other disease that can cause cognitive impairment (e.g., dementia with Lewy bodies, frontotemporal dementia, Parkinson's disease dementia, etc.), intracranial mass impairing cognition, history of traumatic brain injury, normal pressure hydrocephalus, history of clinically significant cerebrovascular disease; b. Excluding other diseases affecting the nervous system, including nervous system infection, epilepsy, and systemic diseases affecting the function of the nervous system; c. Inability to cooperate with cognitive testing; d. Presence of contraindications to MRI examination (e.g., pacemakers, stents, claustrophobia, severe psychiatric symptoms, etc.).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment scale | 1 week pre-suregery and 1 week, 1 month and 3 month after suregery
  ADAS-cog14; range 0 to 90

SECONDARY OUTCOMES:
Alzheimer's Disease Composite Score | 1 week pre-suregery and 1 week, 1 month and 3 month after suregery
  ADCOMS; range 0 to 1.97
Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale for Mild Cognitive Impairment | 1 week pre-suregery and 1 week, 1 month and 3 month after suregery
  Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale for Mild Cognitive Impairment. ADCS-MCI-ADL; range, 0 to 53